CLINICAL TRIAL: NCT03438669
Title: Correlation Between Reading Specific New Visual Acuity Measurement Methods, Patient Self-reported Quality of Life Assessments, Macular Morphological Parameters and Standardized Study Protocol ETDRS Visual Acuity in Wet AMD Patients
Brief Title: Correlation Between Visual Acuity Measurements, Quality of Life and Morphological Parameters in Wet AMD Patients
Acronym: COSP
Status: Completed | Type: Observational
Sponsor: Dr. med. Katja Hatz (Other)
Collaborators: Vista Klinik (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Katja Hatz, Head of Medical Retina Department, Vista Klinik
Organization: Vista Klinik (Other)
Other Study IDs: COSP /EKNZ2016-02216
Record Dates: First submitted 2017-06-09; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Macular Degeneration
Keywords: visual acuity; ETDRS; quality of life
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Patient-reported vision-related quality of life (QOL) outcomes are increasingly incorporated into clinical trials of new treatments for age-related macular degeneration (AMD). In patients with central visual field defects they often do not correlate with distance visual acuity changes as evaluated according to the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Therefore there is the need for better correlated visual acuity (VA) outcome measures for these patients. In a current big trial for treatment of dry AMD (geographic atrophy) reading speed and low luminance visual acuity are used as outcome measures for the first time. However, limited information is available regarding the associations between distance ETDRS visual acuity, reading speed, low luminance visual acuity, contrast sensitivity, morphological parameters and the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) subscales judged relevant to these measures. Evaluating these correlations could provide the basis for objective study outcome parameters which are better correlated to patient-reported outcomes. Further it increases the understanding of the impact of visual impairment on activities and functioning in patients with eye diseases.

There is an immediate benefit to the study patients, as they might gain information regarding their individual results regarding objective VA measures, contrast sensitivity (and their impact on reading ability). Furthermore, the results of the study could be beneficial for future patients due to, e.g., a better understanding of the disease, especially regarding factors which have an impact on their near vision ability and therefore their quality of life. The study could provide a basis to find and include outcome measures which are correlated better with quality of life than ETDRS distance VA for further AMD trials.

DETAILED DESCRIPTION:
3.1 Background and Rationale AGE-RELATED MACULAR Degeneration (AMD) is the leading cause of blindness among European descended people older than 65 years.

Today, the average life expectancy in developed nations is over 80 years and climbing. And yet, the quality of life during those additional years is often significantly diminished by the effects of age-related, degenerative diseases, including age-related macular degeneration (AMD) Central-field loss (CFL) is often a consequence of macular degeneration, necessitating the use of peripheral vision for reading That means that AMD affects the central vision, resulting in central scotomas and therefore the patients have problems with near distance activities like reading while the peripheral visual field is kept preserved.

AMD is a gradually progressive disease that evolves through stages into severe central vision loss. The earliest signs of AMD involve the appearance of extracellular deposits (drusen), sub-retinal deposits of oxidized lipids and proteins beneath the retinal pigment epithelium (RPE), and variable amounts of visible clumps of pigment in the macula. In the intermediate stages of AMD, drusen become larger and pigmentary changes are more severe. In the advanced stages, patients develop either sub-retinal choroidal neovascularization (the exudative or "wet" form of AMD) or the non-neovascular "dry" form of AMD. The dry form of AMD is characterized by sharply demarcated uni- or multi-focal regions of dysfunctional macula, termed geographic atrophy (GA). The GA patches gradually enlarge to involve the RPE and the corresponding neurosensory retina and choriocapillaris layer of the choroid. These progressive and irreversible changes ultimately cause permanent loss of central (macular) vision.

Geographic atrophy (GA) may cause significant compromise of visual function, even when there still is good visual acuity (VA), because of parafoveal scotomas and foveal function abnormalities antedating visible atrophy AMD is a multifactorial disease with largely unknown pathophysiology. It is believed to be caused by cumulative damage over a lifetime leading to progressive deterioration of the RPE, Bruch's membrane and Choriocapillaris-choroid complex (key players in maintaining retinal function), followed by photoreceptor cells damage. However, the locus of primary damage still remains unclear. Identified pathogenic mechanisms to date include a range of genetic and environmental factors related to primary RPE senescence, oxidative stress, alterations in the complement pathway, increased inflammation, changes in the balance of growth factors, and excessive lipofuscin accumulation. Areas of GA are associated with absolute scotomas. Thus, for a period of years, many patients with GA have good VA because of foveal preservation but are limited by the scotomas surrounding the fovea. For example, a patient may have VA of 20/40 or better, but be unable to fit more than a few letters of a word or a full face in the seeing foveal region .Often multiple central scotomas with very small islands of preserved VA, allow the patient to read single optotypes but not the whole word Visual acuity is the most widely used measure of macular function in clinical trials and clinical practice. However, reading ability is an important component of vision function. Reading difﬁculty diminishes quality of life . Improvement in reading performance is one of the main objectives for elderly low-vision patients ETDRS often does not reflect the reading problems of the patient which are essential in daily life. High contrast distance acuity is not the only relevant measure of visual function in relation to the perceived visual performance of a patient with macular disease (Hazel et al. 2000).

The visual impairment experienced by many patients with age-related macular degeneration (AMD) has been found to affect their ability to perform usual activities, which cause psychological distress, and limit their participation in social events. PROs of visual function provide a more comprehensive evaluation of the impact of, and the effects of treatment for AMD Progression of dry AMD can be slowed in many patients through dietary supplements while visual loss from wet AMD is treated with intravitreal administration of anti-vascular growth factor Therefore there is the need to find a better outcome parameter. The primary purpose of the study will be to evaluate if there is a correlation between self-reported reading difficulties and new near vision testing instrument results and secondarily to establish how strong self-reported reading difficulties are-correlated to functional and morphological parameters. To also evaluate how strong the standard distance visual acuity measurements (ETDRS) are correlated to further functional and morphological parameters.

The study could provide a basis to find and include outcome measures which are correlated better with quality of life than ETDRS distance VA for further AMD trials.

ELIGIBILITY:
Incl.Crit.

* To be eligible for participation, patients will be required to have a confirmed diagnosis of wet AMD (including early, intermediate and advanced) from an ophthalmologist at the Vista Klinik, Binningen.
* Best-corrected visual acuity letter score of ≥ 49 letters (Snellen equivalent of 20/100 or better) using ETDRS charts at a distance of 4m.
* Sufficiently clear ocular media, adequate pupillary dilation, and fixation to permit quality fundus imaging
* Age: ≥ 55 years ( to 100 years)
* Wet AMD patients with lesions within the central 1mm ETDRS Grid subfield foveal zone. (The patient has to have a lesion within the 1mm central zone in the better eye). Although foveal involvement is required, lesions underneath the Foveola is not necessary. The maximum distance a lesion should be from the central point is 500µm.

Excl. Crit.

* Significant ocular disease, for example, recurrent infectious or inflammatory ocular disease.
* Patients who received treatment for CNV within the previous 4 days or who had an acute illness or a history of neurologic disease or cognitive impairment that would interfere with study requirements will not be eligible
* The research will be conducted in accordance with the tenets of the Declaration of Helsinki. Informed consent will be obtained from all patients before testing. Thus, all patients not signing informed consent will be excluded from the study.

Ages: 55 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Age: ≥ 55 years ( to 100 years)
  * patients will be required to have a confirmed diagnosis of wet AMD (including early, intermediate and advanced) from an ophthalmologist at the Vista Klinik, Binningen.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
The primary analysis will be to evaluate if there is a correlation between NEI-VFQ-25 near distance subscale and reading speed | 2 hours
  Pearson correlation between NEI VFQ-25 (National Eye Institute Visual Function Questionnaire) near visual acuity sub scale score (questions 5,6,7) (maximum score 1, minimum score 6, higher score indicates worse vision related to quality of life)

SECONDARY OUTCOMES:
Correlation between NEI VFQ-25 near visual acuity subscale score and low luminance visual acuity score | 2 hours
  Pearson correlation between NEI VFQ-25 (National Eye Institute Visual Function Questionnaire) near visual acuity sub scale score (maximum score 1, minimum score 6, higher score indicates worse vision related to quality of life) and low luminance visual acuity and (min 0.3LogMAR, max -0.3LogMAR, higher score indicates indicates worse low luminance acuity)
Correlation between NEI VFQ-25 near visual acuity subscale score and contrast sensitivity score | 2 hours
  Pearson correlation between NEI VFQ-25 (National Eye Institute Visual Function Questionnaire) near visual acuity sub scale score (maximum score 1, minimum score 6, higher score indicates worse vision related to quality of life) and contrast sensitivity score(min 0.00,max 2.25, higher score indicates highest/best contrast sensitivity)
Correlation between NEI VFQ-25 near visual acuity subscale score and near visual acuity subscale score | 2 hours
  Pearson correlation between NEI VFQ-25 (National Eye Institute Visual Function Questionnaire) near visual acuity sub scale score (maximum score 1, minimum score 6, higher score indicates worse vision related to quality of life) and ETDRS 4m distance visual acuity score (min 0.3LogMAR, max -0.3LogMAR, higher score indicates indicates worse ETDRS visual acuity)
Correlation between NEI VFQ-25 near visual acuity subscale score and size of hypo-autofluorescent lesions (mm2) at autofluorescence | 2 hours
  Pearson correlation between NEI VFQ-25 (National Eye Institute Visual Function Questionnaire) near visual acuity sub scale score (maximum score 1, minimum score 6, higher score indicates worse vision related to quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Vista Klinik, Binningen, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
no IPD, this is a not interventional study